CLINICAL TRIAL: NCT00933868
Title: Comparison of Magnesium Chloride Infusions Versus Placebo Administered Concomitantly With 100% Oxygen Given to Patients Who Have Residual Muscle Weakness From a Stroke That Occurred Three Months to Four Years Ago
Brief Title: Magnesium Chloride Versus Placebo in Patients Who Have Had a Stroke
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Relox Medical, LLC (Industry)
Responsible Party: Principal Investigator, Bert Spilker, Lead Principal Investigator, Relox Medical, LLC
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RM-R001
Record Dates: First submitted 2009-06-30; First posted 2009-07-07 (Estimated); Last update posted 2012-05-25 (Estimated); Status verified 2010-09

CONDITIONS: Stroke
Keywords: A stroke that occurred three months to four years ago
MeSH Terms: conditions — Stroke | interventions — Magnesium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Magnesium infusion in patients breathing 100% oxygen (Experimental): Patients will be given six infusions over three weeks. Each infusion will last between 4 and 10 minutes. They will then return to clinic in 1,2 and 3 months for the same tests (but no infusions will be given).
  Interventions: Drug: Magnesium Chloride
- Placebo infusion (Placebo Comparator): The patients will receive six placebo infusions after which they will return to clinic at one, two and three months. At the conclusion of the trial those patients who received placebo may elect to receive the active treatment in another (open label) trial that will begin shortly after this one concludes.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Magnesium Chloride — An infusion of magnesium chloride will be given over 4 to 10 minutes in patients breathing 100% oxygen
  Arms: Magnesium infusion in patients breathing 100% oxygen
Drug: Placebo — A saline placebo will be given as an infusion (six infusions over a three week period) in a double blind manner with the active test agent
  Arms: Placebo infusion

SUMMARY:
The purpose of this study is to evaluate the effect of six intravenous (IV) infusions of magnesium chloride versus placebo in patients who have residual muscle weakness from a stroke that occurred three months to four years ago.

DETAILED DESCRIPTION:
The hypothesis being tested is that these six treatments will improve muscle weakness and lead to an improvement in functioning/activities of daily living as measured by the 100-point Barthel index, three months after their last treatment versus their baseline measure, and that the mean difference between the treatment and placebo groups of patients will be at least three points in this index.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects of either sex above 18 years of age
2. Documented history of stroke 3 months to four years ago
3. Subjects may have had two or more strokes
4. Must have residual muscle weakness with a 25% or greater difference in strength between the right and left sides of the body
5. Must be assessed as a 2 or 3 on the Modified Rankin Scale
6. Must have a Barthel score at or below 85

Exclusion Criteria:

1. Any traumatic brain injury or other brain injury apart from stroke
2. Renal insufficiency or renal failure
3. Any medical or physical condition that would interfere with the measurements to be conducted
4. Any physical therapy in a facility outside their home within three days of screening

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2009-04; Primary Completion 2010-05 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Barthel Index | Infusions are given over 3 weeks and subjects are followed-up at 1, 2 and 3 month intervals after the infusions

SECONDARY OUTCOMES:
Improvement in muscle strength and function | Infusions are given over 3 weeks and subjects are followed-up at 1, 2 and 3 month intervals after the infusions
Change in the Mini-mental status examination | Infusions are given over 3 weeks and subjects are followed up at 1,2, and 3 months after the infusions
Change in balance, coordination, range of motion | Infusions are given over 3 weeks and subjects are followed-up at 1, 2 and 3 months after the infusions
Incidence of adverse events and changes in vital signs | Infusions are given over 3 weeks and subjects are followed-up at 1, 2, and 3 months after the infusions

CONTACTS AND LOCATIONS:
Overall Officials: Bert Spilker, PhD, MD, Principal Investigator — President, Bert Spilker & Associates, LLC
Locations (3):
- United States (3):
  - Born Preventive Healthcare Clinic, PC, Grand Rapids, Michigan
  - Schachter Center for Complementary Medicine, Suffern, New York
  - Comprehensive Heart Care Inc., Toledo, Ohio